CLINICAL TRIAL: NCT06823024
Title: An Observational, Prospective Study to Assess the Utility of a Speech-based Machine Learning Algorithm to Predict Treatment Response to Psychiatric Interventions
Brief Title: Assess the Utility of a Speech-based Machine Learning Algorithm to Predict Treatment Response to Psychiatric Interventions
Status: Enrolling by invitation | Type: Observational
Sponsor: Psyrin Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PSYRIN-0005
Record Dates: First submitted 2025-01-12; First posted 2025-02-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Obsessive Compulsive Disorder (OCD); Bipolar Disorders; Major Depressive Disorder; Post-Traumatic Stress Disorder, PTSD; Generalized Anxiety Disorder (GAD)
Keywords: TMS; Spravato; Esketamine; Treatment response; Speech; Artificial Intelligence; Natural Language Processing; Acoustic Analysis; Acoustic Biomarkers; Vocal Biomarkers; Machine Learning; Mental Health; Speech Analysis
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Bipolar Disorder; Depressive Disorder, Major; Combat Disorders; Generalized Anxiety Disorder; Speech; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Audio of speech collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants prescribed esketamine: Participants who in their normal course of treatment are prescribed and are administered Spravato (esketamine) within 4 weeks of baseline assessment.
- Participants prescribed TMS: Participants who in their normal course of treatment are prescribed and are administered repetitive transcranial magnetic stimulation within 4 weeks of baseline assessment.

SUMMARY:
This is a research study looking at whether the way people speak can help predict how well they'll respond to certain mental health treatments.

The Main Goal:

The researchers want to see if computer analysis of a person's speech patterns can predict whether they'll respond well to two specific treatments: TMS (Transcranial Magnetic Stimulation) and Spravato (a nasal spray medication). They're focusing on people with depression, bipolar disorder, OCD, anxiety, and PTSD.

How It Works:

200 people with these conditions will participate in the study.Participants will record themselves speaking for about 12 minutes, responding to six different prompts.They'll do these recordings before treatment starts, daily during treatment, right after treatment ends, and again four weeks later. Doctors will track how well people are doing using various questionnaires and rating scales The researchers will look for connections between speech patterns and treatment success. The study will last 12 months.

What Makes Someone a "Treatment Success":

The study considers treatment successful if a person's symptoms improve significantly (specifically, a 2-point or greater reduction on a clinical rating scale (called Clinical Global Impression) and stays improved during the follow-up period (4-weeks).

Why This Matters:

If successful, this research could lead to a simple, non-invasive way to help doctors predict which treatments might work best for different patients. This could help people get the most effective treatment more quickly and help healthcare providers use their resources more efficiently.

Safety Consideration The researchers will also check whether doing the speech assessments causes any distress to participants, making sure the evaluation process itself is safe and comfortable.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient status
2. Men and women aged 18-68 years
3. Capable and willing to provide informed consent
4. Able to adhere to the treatment schedule
5. Stable on medication for at least 2 months with no anticipated changes during the study period
6. Diagnosis of MDD, PTSD, or BD
7. Eligible for and scheduled to receive TMS or Spravato (esketamine) treatment to alleviate symptoms of MDD, PTSD, GAD, OCD or BD
8. Fluent in English
9. Access to a stable internet connection and an electronic device with a microphone for voice recording

Exclusion Criteria:

1. Use of any investigational drug within four weeks of the baseline visit
2. If participating in psychotherapy, the patient must have been in stable treatment for at least three months before study entry, with no anticipated changes in the frequency of therapeutic sessions or therapeutic focus during the TMS or Spravato treatment.
3. Intoxication during speech assessments
4. Cognitive impairment that would interfere with study participation or data quality
5. Lack of fluency in English

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll 200 patients diagnosed with Major Depressive Disorder (MDD), Post-Traumatic Stress Disorder (PTSD), or Bipolar Disorder (BD) who are undergoing repetitive Transcranial Magnetic Stimulation (TMS) or Spravato (esketamine) treatment. Participants will represent diverse racial, ethnic, and gender categories, with ages ranging from 18 to 68 years. The eligibility criteria have been designed to capture a wide range of patients, maintaining high ecological validity and ensuring diverse samples.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Treatment response | Change between Baseline and Week 0 (post-intervention)
  ≥ 2 points symptom severity reduction between baseline and after-treatment evaluation on the clinical global impression severity scale (CGI-S) (between 1, normal, not at all ill, and 7, among the most extremely ill patients).

SECONDARY OUTCOMES:
Remission | Change between Baseline and Week 0 (post-intervention), Week 4 (post-intervention)
  Symptoms below the threshold for having the disorder according to CGI-S and clinical judgement.
Stability of treatment response | Change between Baseline and Week 4 (post-intervention)
  ≥ 2 points symptom severity reduction between baseline and follow-up evaluation after-treatment on the clinical global impression severity scale (CGI-S) (between 1, normal, not at all ill, and 7, among the most extremely ill patients).
Distress caused by the online speech assessment | Week 4
  Self-reported distress caused by the online speech assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Julianna Olah, B.Sc., M.A., M.Sc., Ph.D., Study Director — Psyrin Inc.
Locations (2):
- United States (2):
  - Acacia Clinics, Sunnyvale, California
  - Fermata Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided